CLINICAL TRIAL: NCT02960711
Title: Randomized Controlled Trial of Metformin and Dietary Restriction to Prevent Age-related Morbid Events in People With Metabolic Syndrome
Brief Title: Metformin and Dietary Restriction to Prevent Age-related Morbid Events in People With Metabolic Syndrome
Acronym: MeMeMe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: INT 85-13
Record Dates: First submitted 2016-10-21; First posted 2016-11-10 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Metformin; Tablets; Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- METFORMIN (1700MG/DAY) + LIFESTYLE (Experimental): METFORMIN: 2 tablets per day, one at breakfast (or lunch) and one at dinner, of either metformin (two 850 mg tablets/day) + participation in the life-style intervention activities
  Interventions: Drug: Metformin Hydrochloride 850 MG Oral Tablet [Glucophage]
- PLACEBO+ LIFESTYLE (Placebo Comparator): Placebo: (two identical tablets) according to the blind assignment + participation in the life-style intervention activities
  Interventions: Drug: Ludipress, mg stereate, micronized hydrated silica, talcum
- METFORMIN (1700 mg/day) alone (Experimental): METFORMIN: 2 tablets per day, one at breakfast (or lunch) and one at dinner, of either metformin (two 850 mg tablets/day)
  Interventions: Drug: Metformin Hydrochloride 850 MG Oral Tablet [Glucophage]
- PLACEBO alone (Placebo Comparator): Placebo: (two identical tablets) according to the blind assignment
  Interventions: Drug: Ludipress, mg stereate, micronized hydrated silica, talcum

INTERVENTIONS:
Drug: Metformin Hydrochloride 850 MG Oral Tablet [Glucophage]
  Arms: METFORMIN (1700 mg/day) alone; METFORMIN (1700MG/DAY) + LIFESTYLE
Drug: Ludipress, mg stereate, micronized hydrated silica, talcum — Tablet
  Arms: PLACEBO alone; PLACEBO+ LIFESTYLE

SUMMARY:
Phase III randomized controlled trial on men and women with Metabolic syndrome (MetS) to test the hypothesis that comprehensive life-style changes and/or metformin treatment prevent age-related chronic non-communicable diseases (ArCD).

The aim of the present study is to evaluate the effect of a comprehensive life-style intervention (including moderate physical activity and Mediterranean/macrobiotic diet with moderate calorie and protein restriction), and of treatment with Metformin (a calorie restriction mimetic drug) for the prevention of ArCD.

DETAILED DESCRIPTION:
Phase III randomized controlled trial on men and women with MetS to test the hypothesis that comprehensive life-style changes and/or metformin treatment prevent ArCD.

Design:

2x2 factorial: 2,000 volunteers will be randomized in four equal groups of 500 each, and allocated to the following treatments: METFORMIN (1700MG/DAY) + ACTIVE LIFESTYLE INTERVENTION PLACEBO + ACTIVE LIFESTYLE INTERVENTION METFORMIN (1700 mg/day) alone PLACEBO alone The metformin /placebo component of the study will be double blind.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-74, waist circumference equal or greater than 85 cm for women and 100 cm for men, plus at least two other factors among those defining the MetS

Exclusion Criteria:

* Diagnosed diabetes (or baseline fasting glycemia above 7mmol/L at baseline examination)
* Cancer (except skin carcinoma) diagnosed in the last 5 years, or under treatment
* Excessive frailty: in absence of agreed-upon measurements parameters and cutoff points, the investigator will exclude subjects under the lower 5th percentile of the muscular mass distribution estimated by impedance in previous studies
* Conditions that contraindicate the use of MET because might favour lactic acidosis:

  * Renal, cardiac, hepatic, or respiratory insufficiency
  * Serum creatinine <124μmol/L, or proteinuria at baseline examination
  * Current treatment with K-sparing diuretics, or with proton pump inhibitors
  * Excessive alcohol consumption
* Distressing side effects of MET treatment. Nausea and diarrhoea typically occur in about one third of patients receiving MET for the first time at full dose. To avoid dropouts for gastrointestinal discomfort we will treat all volunteers with half the planned dose for one month in order to exclude intolerant subjects before randomization. Participants randomized in the intervention group will continue to take half a dose for one month and then shift to the full dose.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2014-02; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Total incidence of age related chronic diseases | 5 years
  We will retrieve records for all Age related chronic diseases but we will first concentrate the analysis on cancer, coronary heart disease, stroke, and diabetes

SECONDARY OUTCOMES:
Effect of the intervention on total mortality and on the incidence of specific chronic diseases. | 8-10 years
  The measure is a composite outcome measure consisting of multiple measures (results to be reported as a single value for each Arm/Group).
  The outcome measure describes multiple assessments with potentially different Units of Measure as indicated:
  Waist circumference: cm Glycemia: mg/dL Blood pressure: mmHg Total cholesterol, HDL cholesterol: mg/dL Triglycerides: mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Franco Berrino, MD, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baldassari I, Oliverio A, Krogh V, Bruno E, Gargano G, Cortellini M, Casagrande A, Di Mauro MG, Venturelli E, Del Sette Cerulli D, Manuela B, Berrino F, Pasanisi P. Recruitment in randomized clinical trials: The MeMeMe experience. PLoS One. 2022 Mar 25;17(3):e0265495. doi: 10.1371/journal.pone.0265495. eCollection 2022. PMID 35333878
- [Derived] Cortellini M, Casagrande A, Fornaciari G, Del Sette D, Gargano G, Di Mauro MG, Saibene G, Bruno E, Villarini A, Venturelli E, Berrino F, Baldassari I, Oliverio A, Pasanisi P. A management system for randomized clinical trials: A novel way to supply medication. PLoS One. 2019 Feb 22;14(2):e0212475. doi: 10.1371/journal.pone.0212475. eCollection 2019. PMID 30794607
- [Derived] Cortellini M, Berrino F, Pasanisi P. "Open mesh" or "strictly selected population" recruitment? The experience of the randomized controlled MeMeMe trial. Patient Prefer Adherence. 2017 Jul 6;11:1127-1132. doi: 10.2147/PPA.S135412. eCollection 2017. PMID 28740367
- [Derived] Pasanisi P, Gargano G, Gaetana Di Mauro M, Cortellini M, Casagrande A, Villarini A, Bruno E, Roveda E, Saibene G, Venturelli E, Berrino F. A randomized controlled trial of Mediterranean diet and metformin to prevent age-related diseases in people with metabolic syndrome. Tumori. 2018 Mar-Apr;104(2):137-142. doi: 10.5301/tj.5000599. Epub 2018 May 8. PMID 28106245